CLINICAL TRIAL: NCT00003220
Title: Phase II Study of Bryostatin 1 in Patients With Metastatic Colo-Rectal Adenocarcinoma
Brief Title: Bryostatin 1 in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066081; P30CA022453 (NIH); WSU-D-1457; NCI-T97-0065
Record Dates: First submitted 1999-11-01; First posted 2004-08-13 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — bryostatin 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bryostatin 1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of bryostatin 1 in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of bryostatin 1 administered as a 24 hour intravenous infusion every week for 3 weeks during a 4 week course of therapy in patients with colorectal cancer. II. Determine the response duration, time to progression, and survival time in this patient population. III. Determine the qualitative and quantitative toxic effects of bryostatin 1 on this schedule in this patient population.

OUTLINE: Patients are treated with bryostatin 1 as a 24 hour continuous intravenous infusion weekly for 3 weeks followed by 1 week of rest. Courses are repeated every 4 weeks in the absence of unacceptable toxicity or disease progression. Patients who have no toxic effects after the completion of the first course of therapy may have the dose of bryostatin 1 escalated by 1 dose level in subsequent courses. Patients are followed for response duration and time to treatment failure.

PROJECTED ACCRUAL: A total of 13-26 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed colorectal cancer Unresectable disease Measurable disease No uncontrolled brain metastases

PATIENT CHARACTERISTICS: Age: Any age Performance status: SWOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) AST no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: No active infection Not pregnant or nursing Negative pregnancy test for premenopausal women Fertile patients must use effective contraception No concurrent uncontrolled systemic disorders No prior malignant disease within the past year except in situ carcinoma of the cervix or curatively treated basal cell carcinoma of the skin No history of allergy to bryostatin 1 or its vehicle

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: Only one prior chemotherapy regimen in the adjuvant or metastatic setting allowed At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas) No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy (except contraceptives, appetite stimulants and replacement steroids) Radiotherapy: At least 3 weeks since prior radiotherapy No concurrent radiation therapy No concurrent palliative radiation therapy to only site of measurable disease Surgery: Not specified Other: At least 1 month since prior use of any other investigational agent No concurrent use of experimental medications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-02; Primary Completion 2000-11 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A. Philip, MD, PhD, FRCP, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan